CLINICAL TRIAL: NCT01546077
Title: Comparison of Techniques for Placement of Perineural Catheters in the Popliteal Region
Brief Title: Placement of Perineural Catheters in the Popliteal Region
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Sidiropoulou Tatiana, Lecturer in Anesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLOCSTIM1
Record Dates: First submitted 2012-02-03; First posted 2012-03-07 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Foot Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Hydrolocalization technique group (Active Comparator): Technique of placement of popliteal perineural catheter using the hydrolocalization technique with ultrasound
  Interventions: Procedure: Placement of perineural catheters with Hydrolocalization technique using
- Stimulating Catheter technique group (Active Comparator): A technique for placement of popliteal catheter with the aid of a neurostimulator
  Interventions: Procedure: Placement of perineural catheters with Hydrolocalization technique using

INTERVENTIONS:
Procedure: Placement of perineural catheters with Hydrolocalization technique using — Placement of perineural catheters in the popliteal region comparing two techniques. while the drugs used are the same (ropivacaine 0.6% for initial bolus and 0.2% for continuous technique) we will compare dosage required in each group

SUMMARY:
The purpose of this study is to assess the efficacy of the hydrolocalization technique for placement of popliteal perineural catheters in comparison with the stimulating catheters. A non inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* adults
* BMI less than 30

Exclusion Criteria:

* known allergies to local anesthetics or other drugs used
* patient refusal
* any local or systemic contraindication to the use of popliteal block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
consumption of local anesthetics | 36 hours PO

SECONDARY OUTCOMES:
pain scores | 36 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana F Sidiropoulou, MD, PhD, Principal Investigator — Attikon Hospital; Theodosios Saranteas, MD, PhD, Principal Investigator — Attikon Hospital; Georgia G Kostopanagiotou, MD, PhD, Study Chair — Attikon Hospital
Locations (2):
- Attikon Hospital, Athens, Greece
- Policlinico Tor Vergata, Rome, Italy

REFERENCES:
- [Background] Saranteas T, Adoni A, Sidiropoulou T, Paraskeuopoulos T, Kostopanagiotou G. Combined ultrasound imaging and hydrolocalization technique for accurate placement of perineural catheters. Br J Anaesth. 2011 Dec;107(6):1008-9. doi: 10.1093/bja/aer375. No abstract available. PMID 22088876